CLINICAL TRIAL: NCT02701023
Title: Individual Patient Expanded Access - MitoGel for Upper Urinary Tract Urothelial Carcinoma
Brief Title: Compassionate Use of MitoGel in Upper Tract Urothelial Carcinoma
Status: No longer available | Type: Expanded Access
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-000080
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Urothelial Carcinoma Ureteral Location

INTERVENTIONS:
Drug: MitoGel — The patient would then undergo instillation of MitoGel into the affected kidney. The catheter would be left indwelling in the ureter and would be externalized through a urethral catheter. The ureteral and urethral catheters would remain indwelling for the duration of the 6 treatments, which would occur twice weekly for 3 weeks. Following the final instillation, the catheters would be removed. The patient would then undergo ureteroscopic evaluation at 3 months following the final instillation of MitoGel. The total duration of study would be 3 months.

SUMMARY:
The aim of this study is to evaluate the feasibility, safety, and efficacy of MitoGel in the treatment of UTUC in a human subject with low-grade UTUC which is endoscopically unresectable or rapidly recurring, and in whom nephrectomy would likely result in the need for permanent hemodialysis. The study drug would be obtained under the single patient access program approved by the FDA. The patient would then undergo instillation of MitoGel into the affected kidney. The catheter would be left indwelling in the ureter and would be externalized. The ureteral and urethral catheters would remain indwelling for the duration of the 6 treatments, which would occur twice weekly for 3 weeks or once weekly for 6 weeks. Following the final instillation, the catheters would be removed. The patient would then undergo ureteroscopic evaluation at 3 months following the final instillation of MitoGel. The total duration of study would be 3 months. The total number of study patients is 1.

DETAILED DESCRIPTION:
Upper urinary tract urothelial carcinoma (UTUC) is a rare malignant neoplasm arising from the urothelial lining of the renal collecting system and ureters. The current treatment paradigm for UTUC involves endoscopic resection, when technically feasible and oncologically sound, or complete resection of the kidney and ureter (nephroureterectomy) in cases in which organ-sparing treatment is not feasible.

Both organ-sparing and complete resection options present significant technical and clinical challenges. For patients with bilateral disease, an anatomic or functionally solitary kidney, or significant underlying medicorenal disease, treatment with nephroureterectomy would result dialysis dependence, a state which carries with it a significant risk of 5-year mortality in the often elderly and co-morbid patient population affected by UTUC.

MitoGel is a novel investigational product composed of RTGel, a unique hydrogel polymer which exists as liquid at cold temperatures and a viscous gel at body temperatures, and Mitomycin C, a clinically proven safe and effective treatment for urothelial carcinoma in the bladder. MitoGel can be instilled into the upper urinary tract as a cold liquid, where it solidifies to a gel upon warming to body temperature. The agent remains in the upper tract for a period of 4-6 hours, resulting in sustained contact between the tissues and Mitomycin C. Preclinical studies of MitoGel in the Yorkshire swine have demonstrated that both single and serial instillations into the pelvicalyceal system via both retrograde and antegrade approaches are safe, with no observable adverse clinical, laboratory, or histological effects. For these reasons, MitoGel has generated interest as a treatment for UTUC.

For patients with UTUC in whom nephroureterectomy would result in dialysis dependence, and in whom the disease is difficult to manage endoscopically, there is no currently available means to effectively deliver adjuvant chemotherapy to the upper tracts. These patients are thus either condemned to treatment with complete resection of their kidney and resultant hemodialysis, or risk progression of disease to an incurable and unmanageable state. MitoGel represents a promising treatment option for patients who have no other therapeutic options. For these reasons, MitoGel has been granted Orphan Designation Status by the FDA. While clinical trials of MitoGel are currently being planned, no trials are open to date.

The aim of this study is to evaluate the feasibility, safety, and efficacy of MitoGel in the treatment of UTUC in a human subject with low-grade UTUC which is endoscopically unresectable or rapidly recurring, and in whom nephrectomy would likely result in the need for permanent hemodialysis. The study drug would be obtained under the single patient access program approved by the FDA. The patient would then undergo instillation of MitoGel into the affected kidney. The catheter would be left indwelling in the ureter and would be externalized through a urethral catheter. The ureteral and urethral catheters would remain indwelling for the duration of the 6 treatments, which would occur twice weekly for 3 weeks. Following the final instillation, the catheters would be removed. The patient would then undergo ureteroscopic evaluation at 3 months following the final instillation of MitoGel. The total duration of study would be 3 months. The total number of study patients is 1.

ELIGIBILITY:
Inclusion criteria:

* Therapy to be utilized as part of the FDA Compassionate use IND
* Histologically confirmed low grade upper tract urothelial carcinoma which is high-volume and difficult to control using standard ablative therapies
* Anatomically solitary kidney or renal insufficiency significant enough such that nephroureterectomy would result in dialysis dependence
* Willing to consent and participate in a single-patient expanded access use under an FDA IND agreement
* Willing to maintain an indwelling foley catheter for a period of 3 weeks

Exclusion criteria

* Hypersensitivity to mitomycin C or any of the other drug components
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has an active urinary tract infection
* Is unable to tolerate the treatments
* Demonstrates progressively worsening renal dysfunction
* Has a known additional malignancy that is progressing or requires active treatment
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial

Ages: 76 Years to 77 Years | Sex: Male
Age Groups: Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States